CLINICAL TRIAL: NCT06728410
Title: A Phase II Study of Pemigatinib Plus Durvalumab (MEDI4736) in Previously Treated Advanced Intrahepatic Cholangiocarcinoma Patients With FGFR-2 Fusion or Rearrangement
Brief Title: A Phase II Study of Pemigatinib Plus Durvalumab in Previously Treated Advanced Intrahepatic Cholangiocarcinoma Patients With FGFR-2 Fusion or Rearrangement
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mehmet Akce (Other)
Collaborators: AstraZeneca (Industry); Incyte Corporation (Industry); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor-Investigator, Mehmet Akce, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN-GI23-621
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Intrahepatic Cholangiocarcinoma; FGFR2 Gene Rearrangement; FGFR2 Gene Mutation
MeSH Terms: conditions — Cholangiocarcinoma | interventions — pemigatinib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pemigatinib + Durvalumab (Experimental): Pemigatinib 13.5 mg will be taken orally at the same time each day for 14 days (Day 1 through Day 14), followed by 7 days off treatment (Day 15 through Day 21) of each 21 day cycle. Durvalumab 1500 mg IV will be administered every 3 weeks on Day 1 of each 21-day cycle.
  Interventions: Drug: Pemigatinib; Drug: Durvalumab

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib 13.5 mg
  Other Names: PEMAZYRE
Drug: Durvalumab — Durvalumab 1500 mg IV
  Other Names: Imfinzi

SUMMARY:
This is a single arm phase II study of pemigatinib and durvalumab combination in patients with FGFR-2 fusion or rearrangement positive intrahepatic cholangiocarcinoma. Each cycle will be 3 weeks. Pemigatinib is administered at 13.5 mg orally daily 2 weeks on and 1 week off. Durvalumab is administered at 1500 mg intravenously once every 3 weeks. Subjects will require a visit with appropriate laboratory work prior to the start of each cycle. Disease assessment will occur every 9 weeks. Subjects will continue treatment until progression per RECIST 1.1, toxicity or subject/physician decision. A maximum of 24 months (about 35 cycles) of pemigatinib and durvalumab treatment from Cycle 1 Day 1 is allowed.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. ECOG Performance Status of 0 or 1 within 7 days prior to Cycle 1 Day 1.
4. Body weight of > 30 kg.
5. Histologically diagnosed locally advanced unresectable or metastatic intrahepatic cholangiocarcinoma with FGFR-2 fusion or rearrangement detected by Clinical Laboratory Improvement Act (CLIA)-certified assays including commercial tests (Foundation Medicine, Caris, Tempus, Guardant 360 or other platforms of next generation sequencing will be allowed). AJCC, 8th edition. Subjects with gallbladder cancer or ampulla of Vater carcinoma are not eligible.
6. Measurable disease according to RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. Have received gemcitabine cisplatin and durvalumab or another anti-PD-1 Ab for unresectable locally advanced or metastatic cholangiocarcinoma with either disease progression, intolerance to cytotoxic chemotherapy, or have received at least 6 months of therapy with stable disease or partial response. Prior neoadjuvant or adjuvant therapy is permitted if documented disease recurrence occurred ≥ 6 months after the last date of neoadjuvant or adjuvant therapy.
8. Demonstrate adequate organ function as defined below. All screening labs to be obtained within 28 days prior to registration.

   * Absolute Neutrophil Count (ANC): ≥1500/µL
   * Hemoglobin (Hgb): ≥ 9 g/dL; Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
   * Platelet (PLT): ≥ 100 000/µL
   * Calculated creatinine clearance: >40 mL/min
   * Bilirubin: ≤ 1.5 × upper limit of normal (ULN) This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with the sponsor-investigator.
   * Aspartate aminotransferase (AST): ≤ 2.5 × institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
   * Alanine aminotransferase (ALT): ≤ 2.5 × institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
   * International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT): ≤ 1.5 × ULN unless subject is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
9. Females of childbearing potential must have a negative serum pregnancy test at screening.
10. Females of childbearing potential who are sexually active with a male able to father a child must be willing to use an effective method(s) of contraception. Males able to father a child who are sexually active with female of childbearing potential must be willing to use an effective method(s) of contraception.
11. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
12. Must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Prior therapy with a FGFR inhibitor.
2. Current evidence of clinically significant corneal (including but not limited to bullous/band keratopathy, corneal abrasion, inflammation/ulceration, and keratoconjunctivitis) or retinal disorder (including but not limited to macular/retinal degeneration, diabetic retinopathy, and retinal detachment) as confirmed by ophthalmologic examination
3. History of calcium and phosphate homeostasis disorder or systemic mineral imbalance with ectopic calcification of soft tissues (exception: commonly observed calcifications in soft tissues such as the skin, kidney tendon, or vessels due to injury, disease, or aging in the absence of systemic mineral imbalance)
4. Use of any potent CYP3A4 inhibitors or inducers or moderate CYP3A4 inducers within 14 days or 5 half-lives (whichever is longer) before the first dose of study drug. Moderate CYP3A4 inhibitors are not prohibited but should be avoided.
5. History of hypovitaminosis D requiring supraphysiologic doses (eg, 50,000 UI/weekly) to replenish the deficiency. Vitamin D supplements are allowed.
6. Participation in another clinical study with an investigational product during the last 3 months
7. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
8. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤ 28 days prior to the first dose of study regimen. If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by sponsor-investigator.
9. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

   * Patients with Grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the sponsor-investigator.
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with the study regimen may be included only after consultation with the sponsor-investigator.
10. Any concurrent chemotherapy, study drug, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
11. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study regimen.
12. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study regimen. NOTE: Local surgery of isolated lesions for palliative intent is acceptable.
13. History of allogenic organ transplantation.
14. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the sponsor-investigator
    * Patients with celiac disease controlled by diet alone
15. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
16. History of another primary malignancy except for

    * Malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of the study regimen and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
17. History of leptomeningeal carcinomatosis
18. Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry. Has untreated central nervous system (CNS) metastases and/or carcinomatous meningitis identified either on the baseline brain imaging obtained during the screening period or identified prior to signing the ICF. Patients whose brain metastases have been treated may participate provided they show radiographic stability (defined as 2 brain images, both of which are obtained after treatment to the brain metastases. These imaging scans should both be obtained at least four weeks apart and show no evidence of intracranial progression). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either, without the use of steroids, or are stable on a steroid dose of ≤ 10mg/day of prednisone or its equivalent and anticonvulsants for at least 14 days prior to the start of treatment. Brain metastases will not be recorded as RECIST Target Lesions at baseline.
19. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).
20. History of active primary immunodeficiency
21. Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of antiHBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.

    * Participants co-infected with HBV and HCV, or co-infected with HBV and HDV, namely: HBV positive (presence of HBsAg and/or anti HBcAb with detectable HBV DNA); AND
    * HCV positive (presence of anti-HCV antibodies); OR
    * HDV positive (presence of anti-HDV antibodies).
22. Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies).
23. Active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
24. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
25. Receipt of live attenuated vaccine within 30 days prior to the first dose of study regimen. NOTE: Patients, if enrolled, should not receive live vaccine whilst receiving study regimen and up to 90 days after the last dose of study regimen.
26. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control.
27. Known allergy or hypersensitivity to any of the study regimen medications or any of the study regimen medication excipients.
28. Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
29. Patients who have received prior anti-PD-1, anti PD-L1:

    * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
    * All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
    * Must not have experienced a ≥ Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Patients with endocrine AE of ≤ Grade 2 are permitted to enrol if they are stably maintained on appropriate replacement therapy and are asymptomatic.
    * Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
30. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Confirmed objective response rate (ORR) | 24 months
  ORR will include confirmed complete response (CR) + confirmed partial response (PR) and will be determined as per RECIST version 1.1. A confirmed response is defined to be either a CR or PR noted as the objective status on 2 consecutive evaluations at least 4 weeks apart.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 24 months
  PFS is defined as the time from Day 1 of treatment until the criteria for disease progression is met as defined by RECIST version 1.1 or death as a result of any cause.
Disease Control Rate (DCR) | 24 months
  DCR (per RECIST 1.1 as assessed by the Investigator) is defined as the rate of best objective response of CR, PR, or SD according to RECIST 1.1. DCR is defined as the percentage of subjects who have a best objective response of CR or PR or who have SD for at least 9 weeks (±7 days) following the start of study treatment.
Overall Survival | 24 months
  OS is defined as the time from Day 1 of treatment until death from any cause.
Duration of response | 24 months
  DOR (per RECIST 1.1 as assessed by the Investigator) will be defined as the time from the date of first documented response until the first date of documented progression or death in the absence of disease progression (ie, date of PFS event or censoring - date of first response). The end of response should coincide with the date of progression or death from any cause used for the RECIST 1.1 PFS endpoint.
Number of Participants with Adverse Events | 24 months
  Adverse events will be assessed according to the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v5

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Akce, MD, Principal Investigator — Sponsor-Investigator
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No